CLINICAL TRIAL: NCT03411291
Title: The Effect of Statins on Cerebral Blood Flow and Neural Activity-A Non-Randomized Pilot Study
Brief Title: Statins in Cerebral Blood Flow and Neuronal Activity--A Pilot Study
Status: Completed | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Franklin G. Moser, M.D., Director, Neuro-Interventional Imaging; Vice-Chair, Radiology Research, Cedars-Sinai Medical Center
Other Study IDs: CSMC IRB Pro00011194
Record Dates: First submitted 2007-12-26; First posted 2018-01-26 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's, magnetic resonance imaging
MeSH Terms: conditions — Alzheimer Disease | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Diet: MRI/MR Spectroscopy/MR Perfusion: Healthy candidates for statin therapy to lower cholesterol pre-electing to lower cholesterol by diet for three months. Candidates in this arm have pre-elected to lower cholesterol by diet as described under the care of their treating physicians. Candidates will have 1 (one) brain MRI / MR spectroscopy/MR resonance perfusion scan at baseline and 1 (one) brain MRI / MR spectroscopy/MR resonance perfusion scan at 3 (three) months.
- Statin: MRI/MR Spectroscopy/MR Perfusion: Healthy candidates for statin therapy pre-electing to lower their cholesterol using atorvastatin (Lipitor) 20 mg per day as prescribed by their treating physician per standard of care. There are no research-related interventions for this group. Candidates will have 1 (one) brain MRI / MR spectroscopy/MR resonance perfusion scan at baseline and 1 brain MRI / MR spectroscopy/MR resonance perfusion scan at 3 months.
  Interventions: Device: MRI, MR Spectroscopy, MR Perfusion

INTERVENTIONS:
Device: MRI, MR Spectroscopy, MR Perfusion — One brain MRI/MR Spectroscopy/MR Perfusion at baseline and one brain MR/MR Spectroscopy/MR Perfusion at 3 months.
  Groups: Statin: MRI/MR Spectroscopy/MR Perfusion

SUMMARY:
Specific Aim: Demonstrate that statins have an effect on cerebral blood flow and neuronal activity

DETAILED DESCRIPTION:
A number of recent of recent studies suggests that statins, typically used to lower blood cholesterol have an effect on the brain. Patients treated with statins may have increased blood flow in the brain resulting in increased activity of the brain's neurons. The neuronal system is linked to memory. Brain magnetic resonance imaging (MRI) with magnetic resonance spectroscopy (MRS) and magnetic resonance perfusion (MRP) will be used to assess changes in neuronal activity in patients receiving statins vs. patients not receiving statins.

This is a single-site non-randomized pilot study. The study will include twenty (20), healthy consenting patients between the ages of 45 and 65 who are candidates for statin therapy as determined by their cardiologist(s). Two imaging visits will be required, one magnetic resonance imaging with Magnetic Resonance Spectroscopy and Magnetic Resonance Perfusion at baseline and one magnetic resonance imaging with magnetic resonance Spectroscopy and Magnetic Resonance Perfusion three months later as described.

Patients will have selected their course of clinical treatment prior to recruitment. Ten patients will have elected to start statin therapy with Lipitor and ten patients will have elected to initially lower their cholesterol levels with diet, independent of their participation in the study.

Participants on the "statin arm" will receive a dose of 20 mg per day of Lipitor and will receive a baseline brain Magnetic Resonance Imaging with Magnetic Resonance Spectroscopy and Magnetic Resonance Perfusion prior to receiving Lipitor and follow-up brain Magnetic Resonance Imaging with Magnetic Resonance Spectroscopy and Magnetic Resonance Perfusion three months after beginning Lipitor.

Participants on the "diet arm" will receive a baseline brain magnetic resonance imaging with Magnetic Resonance Spectroscopy and Magnetic Resonance Perfusion at the beginning of the study and follow-up brain magnetic resonance imaging with magnetic resonance spectroscopy and magnetic resonance perfusion three months later.

ELIGIBILITY:
Inclusion Criteria:

1. Otherwise healthy adults, male or female
2. Age 45-65,
3. Prior to treatment with any statin at a moderate or high dose -

Exclusion Criteria:

1. Previous cerebral vascular accident,
2. Traumatic brain injury,
3. Subarachnoid hemorrhage,
4. Vascular dementia,
5. Alzheimer's Disease A
6. Any other known vascular pathologies of the brain.
7. Patients taking and/or receiving other known cerebrovascular enhancing medication/herbs and/or treatment (examples: tPA, gingko, triple H therapy, stenting procedures, etc.)
8. Previous neurosurgery or intracranial procedures.
9. Contraindication to MRI (pacemaker, neurostimulator, other surgical implants or metals which would contraindicate MRI).

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 patients male and female
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2007-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
MRI Spectroscopy | 3 months
  Changes in metabolite concentration in areas of the brain linked to memory measured by MR spectroscopy with quantitative post processing
MRI Perfusion | 3 months
  Changes in perfusion in areas of the brain linked to memory measured by DCS perfusion imaging

CONTACTS AND LOCATIONS:
Overall Officials: Franklin G. Moser, M.D., Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, S. Mark Taper Foundation Imaging Center, Los Angeles, California, United States

REFERENCES:
- See also: Article: Amarenco P, Lavallée P & Touboul P-J. (2004) Stroke prevention, blood cholesterol, and statin. Lancet Neurol 3: 271-278. — https://www.ncbi.nlm.nih.gov/pubmed/15099541
- See also: Review: Forsting M. Weber J. MR perfusion imaging: a tool for more than stroke. — https://www.ncbi.nlm.nih.gov/pubmed/15457993
- See also: Article: Brain microvascular changes in Alzheimer's disease and other dementias. — https://www.ncbi.nlm.nih.gov/pubmed/9329677